CLINICAL TRIAL: NCT05482659
Title: The Effect of Online Transtheoretic Model Based Health Education on Overweight University Students on Nutrition and Physical Activity Change Processes.
Brief Title: The Effect of Online Transtheoretic Model Based Health Education on Overweight University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, CANSU YAŞAR, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SaglikBilimleriUniversity
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Public Health Nursing
Keywords: transtheoretical model; Public Health Nursing; University Student

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Health education on healthy nutrition and regular physical activity based on the transtheoretic model was given to overweight university students in the experimental group once a week (every 4 weeks) using the online education method.
  Interventions: Behavioral: Health education on healthy nutrition and regular physical activity based on the transtheoretic model
- control group (No Intervention): No attempt was made to the students in the control group during the intervention process. When the intervention process of the experimental group was finished, the materials used in health education were shared with the students.

INTERVENTIONS:
Behavioral: Health education on healthy nutrition and regular physical activity based on the transtheoretic model — An announcement was made by visiting all the faculties at Nuh Naci Yazgan University, stating the content of the research and the duration of the research. Among the volunteer students, students who met the inclusion criteria were included in the study. Afterwards, the students were assigned to the groups by the statistician using a simple randomization method. As a result of the pre-test, it was determined which change stage each student was in according to the Transtheoretic model (TTM). The students were not given information about which group they were in and what stage they were in according to TTM. Health education was given to university students once a week by online education method and it took 4 weeks-30 days to complete the research. The average duration of the health education given to each student is 30-45 minutes. When the training process was over, the post-test questions were sent to the students by the online survey method.
  Arms: Experimental

SUMMARY:
Aim: In this study, it was aimed to determine the effect of health education given to overweight university students based on the Transtheoretic Model (TTM) on nutrition and physical activity behaviors.

Materials and Methods: The research was conducted in a randomized controlled experimental design. The sample of the study consisted of 54 students, 27 of which were in the experimental group and 27 in the control group, who met the inclusion criteria between October 2021 and November 2021. Students were divided into nutrition and exercise change stages groups according to TTM. The students in the experimental group were given one-on-one health education in accordance with the TTM change stages, using the online method. In the study, data were collected using the Sociodemographic Form, Nutrition and Exercise Stage Determination Form according to TTM, Nutrition Change Processes Scale (NCPS) and Exercise Change Processes Scale (ECPS). Chi-square test and t test for dependent and independent groups were used in the analysis of the data obtained. Statistical significance level was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research,
* University students without chronic diseases
* BMI level between 24.9 and 30,
* Open to communication and cooperation,
* Internet and smartphone/tablet/computer etc. owner.

Exclusion Criteria:

* BMI level of 24.9 and below,
* Using any drug,
* Who left the research voluntarily.
* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Stages of change according to the transtheoretic model - pre-intervention and post-intervention | 4 weeks
  The stages of change of the transtheoretic model were measured before and after the intervention to determine that university students changed their unhealthy diet and insufficient physical activity behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu Yaşar, 1, Principal Investigator — cyasar@nny.edu.tr
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Küme Evler Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No